CLINICAL TRIAL: NCT01648322
Title: A Phase II, Randomized, Multi-Centre, Open-Label, Active-Controlled, Dose-Finding Trial of F-627 in Women With Breast Cancer Receiving Myelotoxic Chemotherapy
Brief Title: Dose-Finding Trial of F-627 in Women With Breast Cancer Receiving Myelotoxic Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EVIVE Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-627-02
Record Dates: First submitted 2012-04-27; First posted 2012-07-24 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer; Neutropenia
Keywords: Breast Cancer; Taxotere Chemotherapy; Neulasta; efficacy and safety; single cycle doses of F-627; pegfilgrastim
MeSH Terms: conditions — Breast Neoplasms; Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 80 µg/kg/dose of F-627 (Experimental): This dose of F-627 given only to subjects that are to have TC chemotherapy.
  Interventions: Drug: F-627
- 240 µg/kg/dose of F-627 (Experimental): This dose of F-627 given to subjects receiving TC or TAC chemotherapy.
  Interventions: Drug: F-627
- 320 µg/kg/dose of F-627 (Experimental): This dose of F-627 given to subjects receiving TC or TAC chemotherapy.
  Interventions: Drug: F-627
- Neulasta® (pegfilgrastim) (Active Comparator): Given to subjects receiving TC or TAC chemotherapy.
  Interventions: Drug: Neulasta® (pegfilgrastim)

INTERVENTIONS:
Drug: F-627 — subcutaneous injection given 1 per chemotherapy.
  Arms: 240 µg/kg/dose of F-627; 320 µg/kg/dose of F-627; 80 µg/kg/dose of F-627
Drug: Neulasta® (pegfilgrastim) — Single dose injection given once per chemotherapy cycle.
  Arms: Neulasta® (pegfilgrastim)

SUMMARY:
This is a randomized open label dose finding study to evaluate the efficacy and safety of F-627 on women with Stage I-IV breast cancer receiving chemotherapy treatment.

DETAILED DESCRIPTION:
This is a randomized, multi-center, dose finding, open label, positive controlled Phase II study of the efficacy and safety of once-per-cycle of F-627 compared with Neulasta® (pegfilgrastim) in women with breast cancer who are receiving myelotoxic chemotherapy (TC: docetaxel + cyclophosphamide or TAC: docetaxel + doxorubicin + cyclophosphamide).

The primary objective of this study is to evaluate the efficacy and safety of various single cycle doses of F-627 as compared with the standard dosing of Neulasta® (pegfilgrastim) in breast cancer patients experiencing myelotoxic chemotherapy. Myelotoxicity in this study will be defined by the duration of moderate neutropenia; the number of days in which the patient has had an absolute neutrophil count (ANC) < 1.0 × 10^9/L during the first cycle of their chemotherapy treatment (each chemotherapy cycle is expected to last 21 days). This, by definition, includes grade 3 (moderate) and grade 4 (severe) neutropenia. Doses of F-627 to be tested for subjects receiving TC chemotherapy are 80 µg/kg/dose, 240 µg/kg/dose, and 320 µg/kg/dose. For subjects receiving TAC chemotherapy, only 240 µg/kg/dose and 320 µg/kg/dose are to be tested.

ELIGIBILITY:
Inclusion Criteria:

* Show evidence of a signed (personally or by a legally acceptable representative) and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial.
* Females ≥ 18 years of age.
* Diagnosed with Stage I-IV breast cancer.
* Subject is scheduled to undergo 4 cycles of TC or TAC chemotherapy (Taxotere®, doxorubicin and cyclophosphamide, 75, 50 and 600 mg/m2, respectively).
* ECOG Performance status of ≤ 2.
* White Blood Cell count (WBC) ≥ 4.0 × 109/L, hemoglobin ≥ 11.5 g/dL and a platelet count ≥ 150 × 109/L.
* Demonstrate adequate renal, hepatic function (Liver function tests (ALT, AST, alkaline phosphatase and total bilirubin)) should be less than 2.5x upper limits of normal (ULN). Serum creatinine should be less than 1.7x ULN.
* All subjects must agree to use at least one of the following types of contraception: intrauterine device, implantable progesterone device, progesterone intramuscular injection, or oral contraceptive, which has been started at least one month prior to visit one and will continue for the duration of the trial. The contraceptive patch or condom use with spermicide are also acceptable forms of contraception as long as they will be used continually throughout the duration of the trial.

Exclusion Criteria:

* Subject is <18 or ≥ 75 years of age.
* Disease progression has occurred while receiving a taxane regimen.
* Subject has undergone radiation therapy within 4 weeks of enrollment.
* Subject has undergone bone marrow or stem-cell transplantation.
* Subject has a history of prior malignancy other than breast cancer.
* Subjects that have used G-CSF within 6 weeks of the screening period are also excluded
* Subject has had chemotherapy within 365 days of screening
* Subject has documented congestive heart failure, cardiomyopathy or myocardial infarction by clinical diagnosis, ECG test, or any other relevant test.
* History of alcohol or drug abuse that would interfere with the ability to be compliant with the study procedure.
* Unwillingness to participate in the study.
* Any underlying medical condition that, in the Investigator's opinion, would make the administration of study drug hazardous to the patient or that would obscure the interpretation of adverse events.
* Receiving other investigational drugs or biologics within 1 month or five half lives of enrollment.
* Any condition, which can cause splenomegaly.
* Chronic constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease.
* ALT, AST, alkaline phosphatase > 2.5 upper limit of normal.
* Patients with active infection, or known to be infected with chronic active Hepatitis B within the last 1 year (unless shown at the time of study entry to be Hepatitis B antigen negative), or having any history of Hepatitis C.
* Women who are pregnant or breast-feeding.
* Patients known to be seropositive for HIV, or who have had an AIDS defining illness or a known immunodeficiency disorder.
* Patients with a history of tuberculosis or exposure to tuberculosis. Patients that have received a prior chest X-ray for suspicion of tuberculosis are also excluded unless they have been confirmed to be PPD negative or they had latent tuberculosis that has been previously treated.
* Subjects with Sickle Cell disease
* Subjects with known hypersensitivity to E.coli derived proteins' pegfilgrastim' filgrastim, or any other component of the study drug.

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Community Hospital of Anderson, Anderson, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glaspy J, Bondarenko I, Krasnozhon D, Rutty D, Chen J, Fu Y, Wang S, Hou Q, Li S. Efbemalenograstim alfa not inferior to pegfilgrastim in providing neutrophil support in women with breast cancer undergoing myelotoxic chemotherapy: results of a phase 2 randomized, multicenter, open-label trial. Support Care Cancer. 2024 Jan 9;32(2):91. doi: 10.1007/s00520-023-08260-x. PMID 38194162

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 80 µg/kg/Dose of F-627 | 240 µg/kg/Dose of F-627 | 320 µg/kg/Dose of F-627 | Neulasta® (Pegfilgrastim)
Started | 35 | 67 | 65 | 65
Completed | 33 | 62 | 60 | 61
Not Completed | 2 | 5 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 80 µg/kg/Dose of F-627 | 240 µg/kg/Dose of F-627 | 320 µg/kg/Dose of F-627 | Neulasta® (Pegfilgrastim) | Total
Number analyzed (Participants) | 35 | 67 | 65 | 65 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (10.3) | 47.9 (10.1) | 48.9 (10.3) | 48.2 (10.9) | 48.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 67 | 65 | 65 | 232
  Male | 0 | 0 | 0 | 0 | 0
weight [Mean (Standard Deviation); unit: kg] | 73.28 (17.12) | 70.89 (14.44) | 70.22 (12.94) | 71.28 (14.09) | 71.18 (14.32)
Height [Mean (Standard Deviation); unit: cm] | 164.88 (5.66) | 163.58 (8.15) | 162.90 (5.66) | 162.80 (6.99) | 163.37 (6.83)
ECOG status [Count of Participants; unit: Participants] — The ECOG Scale of Performance Status describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.).
  GRADE 0. Fully active
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all self care but unable to carry out any work activities
  A subject's ECOG grade is determined by the study doctor based on the established criteria listed above.
  Grade 0 is best. Grade 2 is worse than Grade 1.
  Participants
    Grade 0 | 25 | 40 | 42 | 41 | 148
    Grade 1 | 10 | 27 | 23 | 24 | 84
    Grade 2 | 0 | 0 | 0 | 0 | 0
Cancer Stage at screen [Number; unit: participants]
  I | 1 | 12 | 12 | 9 | 34
  II | 25 | 28 | 32 | 31 | 116
  III | 9 | 23 | 18 | 23 | 73
  IV | 0 | 4 | 3 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Duration of Moderate Neurtopenia Post First Chemotherapy Administration
Description: Number of days In which the patient has had an absolute neutrophil count (ANC) Level < 2.0 x 10^9/L after first cycle of chemotherapy
Time Frame: The first of 4, 21 Day Chemotherapy Cycles
Population: per protocol population
Measure: Mean (Standard Deviation); unit: days
Groups:
- 80 µg/kg/Dose of F-627(TC): This dose of F-627 given only to subjects that are to have TC chemotherapy.
  F-627: subcutaneous injection given 1 per chemotherapy.
- 240 µg/kg/Dose of F-627 (TC); 320 µg/kg/Dose of F-627 (TC): This dose of F-627 given to subjects receiving TC or TAC chemotherapy.
  F-627: subcutaneous injection given 1 per chemotherapy.
- Neulasta® (Pegfilgrastim) (TC): Neulasta fixed dose of 6mg given to subjects receiving TC or TAC chemotherapy.
  Neulasta® (pegfilgrastim): Single dose injection given once per chemotherapy cycle.
- 240 µg/kg/Dose of F-627 (TAC); 320 µg/kg/Dose of F-627 (TAC): This dose of F-627 given to subjects receiving TAC chemotherapy.
  F-627: subcutaneous injection given 1 per chemotherapy.
- Neulasta® (Pegfilgrastim) (TAC): Neulasta fixed dose of 6mg given to subjects receiving TAC chemotherapy.
  F-627: subcutaneous injection given 1 per chemotherapy.
Arm/Group | 80 µg/kg/Dose of F-627(TC) | 240 µg/kg/Dose of F-627 (TC) | 320 µg/kg/Dose of F-627 (TC) | Neulasta® (Pegfilgrastim) (TC) | 240 µg/kg/Dose of F-627 (TAC) | 320 µg/kg/Dose of F-627 (TAC) | Neulasta® (Pegfilgrastim) (TAC)
Number analyzed (Participants) | 35 | 37 | 31 | 35 | 30 | 29 | 30
days | 0.6 (1.26) | 0.6 (1.01) | 0.4 (0.75) | 0.3 (0.56) | 2.1 (1.58) | 2.1 (1.46) | 1.8 (1.28)

2. Secondary Outcome: Duration in Days of Grade 3 and Grade 4 Neutropenia for All 4 Chemotherapy Cycles.
Description: Number of days In which the patient has had an ANC < 1.0 × 10^9/L (Grade 3) or ANC < .5 × 10^9/L (Grade 4) post each chemotherapy
Time Frame: Measured for each of the 4, 21 day chemotherapy cycles.
Population: PP population
Measure: Mean (Standard Deviation); unit: Days
Groups:
- 240 µg/kg/Dose of F-627; 320 µg/kg/Dose of F-627: This dose of F-627 given to subjects receiving TC chemotherapy.
  F-627: subcutaneous injection given 1 per chemotherapy.
- Neulasta® (Pegfilgrastim): Given to subjects receiving TC chemotherapy.
  Neulasta® (pegfilgrastim): Single dose injection given once per chemotherapy cycle.
- 240 µg/kg/Dose of F-627- TAC; 320 µg/kg/Dose of F-627 -TAC: This dose of F-627 given to subjects receiving TAC chemotherapy.
  F-627: subcutaneous injection given 1 per chemotherapy.
- Neulasta® (Pegfilgrastim) -TAC: Given to subjects receiving TAC chemotherapy.
  Neulasta® (pegfilgrastim): Single dose injection given once per chemotherapy cycle
Arm/Group | 80 µg/kg/Dose of F-627 | 240 µg/kg/Dose of F-627 | 320 µg/kg/Dose of F-627 | Neulasta® (Pegfilgrastim) | 240 µg/kg/Dose of F-627- TAC | 320 µg/kg/Dose of F-627 -TAC | Neulasta® (Pegfilgrastim) -TAC
Number analyzed (Participants) | 35 | 37 | 31 | 35 | 30 | 29 | 30
Days | 0.4 (0.95) | 0.2 (0.55) | 0.2 (0.54) | 0.1 (0.18) | 1.6 (1.51) | 1.6 (1.17) | 1.2 (1.23)

3. Secondary Outcome: The Incidence Rate of Febrile Neutropenia
Description: The incidence rate of febrile neutropenia for each arm of the study will be recorded for 4 chemotherapy cycles. Each cycle is expected to last 21 Days.
Time Frame: Measured for each of the 4, 21 day chemotherapy cycles.
Population: PP population
Measure: Count of Participants; unit: Participants
Arm/Group | 80 µg/kg/Dose of F-627 | 240 µg/kg/Dose of F-627 | 320 µg/kg/Dose of F-627 | Neulasta® (Pegfilgrastim)
Number analyzed (Participants) | 35 | 67 | 65 | 65
Participants | 0 | 0 | 2 | 2

4. Secondary Outcome: The Duration in Days of Total Grade 2-4 Neutropenia
Description: Number of says in which the patient has had an ANC Level ANC < 1.5 × 109/L) post each chemotherapy
Time Frame: Measured for each of the 4, 21 day chemotherapy cycles.
Population: PP population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 240 µg/kg/Dose of F-627- TAC | 320 µg/kg/Dose of F-627 -TAC | Neulasta® (Pegfilgrastim) -TAC
Number analyzed (Participants) | 30 | 29 | 30
Days | 2.1 (1.48) | 2.0 (1.31) | 1.7 (1.49)

5. Secondary Outcome: The Time to ANC Recovery Post Nadir
Description: The time to ANC recovery post nadir for each patient, for each of their chemotherapy cycles will be recorded; recovery for this protocol is defined as achieving an ANC ≥ 2.0 × 10^9/L after the expected ANC nadir (expected nadir is typically 4-6 days post chemotherapy administration). Each chemotherapy cycle is expected to last 21 days.
Time Frame: Measured for each of the 4, 21 day chemotherapy cycles.
Population: TAC PP population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 240 µg/kg/Dose of F-627- TAC | 320 µg/kg/Dose of F-627 -TAC | Neulasta® (Pegfilgrastim) -TAC
Number analyzed (Participants) | 30 | 29 | 30
Days | 2.4 (1.56) | 2.0 (1.27) | 1.9 (1.20)

6. Secondary Outcome: The Incidence Rates of Grade 2, Grade 3, and Grade 4 Neutropenia for All Chemotherapy Cycles
Description: The incidence rate of mild, moderate and sever neutropenia for each arm of the study will be recorded for 4 chemotherapy cycles. Each cycle is expected to last 21 Days.
Time Frame: Measured for each of the 4, 21 day chemotherapy cycles.
Population: PP population
Measure: Count of Participants; unit: Participants
Arm/Group | 80 µg/kg/Dose of F-627(TC) | 240 µg/kg/Dose of F-627 (TC) | 320 µg/kg/Dose of F-627 (TC) | Neulasta® (Pegfilgrastim) (TC) | 240 µg/kg/Dose of F-627 (TAC) | 320 µg/kg/Dose of F-627 (TAC) | Neulasta® (Pegfilgrastim) (TAC)
Number analyzed (Participants) | 35 | 37 | 31 | 35 | 30 | 29 | 30
Participants | 17 | 14 | 11 | 10 | 28 | 25 | 25

7. Secondary Outcome: The Depth of the ANC Nadir for All Chemotherapy Cycles
Description: The depth of ANC nadir for each cycle is defined as the minimal ANC value for a subject in each chemotherapy cycle. The depth of the ANC nadir for each arm of the study will be recorded for 4 chemotherapy cycles.
Time Frame: Measured for each of the 4, 21 day chemotherapy cycles
Population: PP population
Measure: Mean (Standard Deviation); unit: x 10^9/L
Arm/Group | 80 µg/kg/Dose of F-627(TC) | 240 µg/kg/Dose of F-627 (TC) | 320 µg/kg/Dose of F-627 (TC) | Neulasta® (Pegfilgrastim) (TC) | 240 µg/kg/Dose of F-627 (TAC) | 320 µg/kg/Dose of F-627 (TAC) | Neulasta® (Pegfilgrastim) (TAC)
Number analyzed (Participants) | 35 | 37 | 31 | 35 | 30 | 29 | 30
x 10^9/L
  Cycle 1 | 2.09 (1.5) | 2.41 (1.86) | 3.00 (2.61) | 3.05 (2.31) | 0.68 (1.06) | 0.86 (1.41) | 0.78 (1.28)
  Cycle 2: number analyzed (Participants) | 34 | 35 | 30 | 34 | 27 | 28 | 28
  Cycle 2 | 3.45 (2.54) | 3.74 (2.09) | 4.71 (3.09) | 4.11 (1.59) | 1.87 (1.65) | 1.79 (1.56) | 1.65 (1.30)
  Cycle 3: number analyzed (Participants) | 34 | 34 | 29 | 34 | 27 | 28 | 27
  Cycle 3 | 3.47 (2.18) | 3.80 (2.43) | 4.91 (2.68) | 4.78 (2.36) | 1.41 (1.22) | 1.43 (1.51) | 1.91 (1.37)
  Cycle 4: number analyzed (Participants) | 34 | 34 | 29 | 33 | 25 | 28 | 27
  Cycle 4 | 2.93 (1.74) | 3.56 (2.45) | 4.75 (3.45) | 3.99 (2.46) | 1.35 (1.22) | 1.94 (2.15) | 1.91 (1.46)

ADVERSE EVENTS:
Time Frame: Subjects were to be followed up 30 days after the last study visit for identification of AEs. Subsequent to the 30 day AE follow-up, subjects who discontinued due to FN were to be followed up for an additional 30 days to identify further FN events or severe neutropenia (defined as ANC <0.5×109/L) with duration >2 days. Any Grade 3 or 4 AEs or SAEs were to be followed up until they had resolved or stabilized.
Description: The NCI CTCAE v4.0 grading system was used in AE reporting to provide a standard language to describe toxicities, to facilitate tabulation and analysis of the data, and to facilitate the assessment of the clinical significance of all AEs. AEs were to be recorded and graded 1 to 5 according to the CTCAE grades provided below:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe and undesirable AE Grade 4 Life-threatening or disabling AE Grade 5 Death
Groups:
- Neulasta® (Pegfilgrastim): Neulasta fixed dose of 6mg given to subjects receiving TC or TAC chemotherapy.
  Neulasta® (pegfilgrastim): Single dose injection given once per chemotherapy cycle.
Arm/Group | 80 µg/kg/Dose of F-627 | 240 µg/kg/Dose of F-627 | 320 µg/kg/Dose of F-627 | Neulasta® (Pegfilgrastim)
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/67 | 1/65 | 4/65
Other Adverse Events (participants affected / at risk) | 32/35 | 63/67 | 61/65 | 59/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 80 µg/kg/Dose of F-627 (N=35) | 240 µg/kg/Dose of F-627 (N=67) | 320 µg/kg/Dose of F-627 (N=65) | Neulasta® (Pegfilgrastim) (N=65)
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis Toxic (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 80 µg/kg/Dose of F-627 (N=35) | 240 µg/kg/Dose of F-627 (N=67) | 320 µg/kg/Dose of F-627 (N=65) | Neulasta® (Pegfilgrastim) (N=65)
Alopecia (Skin and subcutaneous tissue disorders) | 27 | 49 | 44 | 52
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4 | 3 | 2
Asthenia (General disorders) | 11 | 13 | 21 | 20
Fatigue (General disorders) | 5 | 13 | 12 | 10
Chest pain (General disorders) | 0 | 2 | 4 | 0
Nausea (Gastrointestinal disorders) | 17 | 22 | 23 | 28
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 4 | 7
Vomiting (Gastrointestinal disorders) | 3 | 0 | 6 | 4
Neutropenia (Blood and lymphatic system disorders) | 6 | 25 | 21 | 17
Leukopenia (Blood and lymphatic system disorders) | 3 | 12 | 8 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 11 | 11 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 1
Headache (Nervous system disorders) | 5 | 5 | 7 | 4
Dizziness (Nervous system disorders) | 3 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4 | 5 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days